CLINICAL TRIAL: NCT00268307
Title: Cellular Transplantation of Autologous Bone Marrow-Derived Stem Cells Following Myocardial Infarction
Brief Title: Bone Marrow Stem Cell Infusion Following a Heart Attack
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Minneapolis Heart Institute Foundation (Other)
Collaborators: Allina Health System (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: Quadruple | Purpose: Treatment
Other Study IDs: opt001
Record Dates: First submitted 2005-12-20; First posted 2005-12-22 (Estimated); Last update posted 2013-12-05 (Estimated); Status verified 2013-12

CONDITIONS: Acute Myocardial Infarction
Keywords: Cell therapy

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (1):
- Cell therapy (Experimental): Intracoronary, one time infusion of autologous, unfractionated bone marrow mononuclear cells.
  Interventions: Drug: Autologous, Unfractionated Bone Marrow Mononuclear Cells

INTERVENTIONS:
Drug: Autologous, Unfractionated Bone Marrow Mononuclear Cells — Intracoronary infusion of Autologous, Unfractionated Bone Marrow Mononuclear Cells. Dose is 100,000,000 cells. One time infusion over 20 minutes.

SUMMARY:
The goal of this study is to determine the safety of giving a patient's own bone marrow-derived stem cells delivered with a catheter (tube) into the coronary arteries (blood vessels of the heart). Stem cells are simple cells produced by the bone marrow that can develop into many types of cells. It is possible that these cells will decrease the size of damage caused to the heart from a heart attack and increase the pumping efficiency of the heart; which can be decreased due to a heart attack. The stem cells will be taken from bone marrow and then given back into the heart vessels.

DETAILED DESCRIPTION:
This protocol will test the hypothesis that an intracoronary infusion of autologous, unfractionated, bone marrow mononuclear cells will attenuate infarct size and improve left-ventricular function in 60 patients following an acute anterior myocardial infarction who have undergone successful revascularization with PTCA/stenting.

ELIGIBILITY:
Inclusion Criteria:

* Patients age at least 21 years of age
* Patients with an acute anterior myocardial infarction limited to the proximal or mid-LAD with an artery diameter of at least 2.5 mm.
* Ability to undergo cell therapy procedure within 2 to 7 days following acute MI and PTCA/stenting.
* Ejection fraction following reperfusion with PTCA/stenting is between 30% and 50% as assessed by left-ventriculography or echocardiography.
* Consent to protocol and agree to comply with all follow-up visits and studies.

Exclusion Criteria:

* History of sustained ventricular arrhythmias not related to their acute myocardial infarction who do not have an ICD.
* Require coronary artery bypass surgery or percutaneous revascularization due to the presence of residual coronary stenosis > 70% luminal obstruction in the non-infarct related vessel.
* History of malignancy within the past 5 years excluding non-melanoma skin cancer or cervical cancer in-situ.
* History of anemia (Hb < 9.0 mg/dl).
* History of thrombocytosis.
* PT or PTT greater than the upper limits of normal.
* Life expectancy less than one year.
* Patients on chronic dialysis.
* History of untreated alcohol or drug abuse.
* Currently enrolled in another Investigational drug or device trial.
* History of stroke or TIA within the past 6 months.
* History of severe valvular heart disease (aortic valve area < 1.0 cm2 or > 3+ mitral regurgitation.
* Pregnancy
* Subjects who are HIV, hepatitis B or C positive.
* Patients with active inflammatory or autoimmune disease on chronic immunosuppressive therapy.
* Contraindications to cardiac MRI

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 41 (Actual)
Dates: Start 2005-12; Primary Completion 2010-01 (Actual); Study Completion 2010-09 (Actual)

PRIMARY OUTCOMES:
Safety as measured by holter monitor, laboratory assessments, and cardiac MRI | 6 months

SECONDARY OUTCOMES:
Improvement of left ventricular function as assessed by serial measurements of infarct size and LV function by cardiac MRI in the active treatment group versus placebo. | 6 months

CONTACTS AND LOCATIONS:
Overall Officials: Jay Traverse, MD, Principal Investigator — Minneapolis Heart Institute
Locations (1):
- Minneapolis Heart Institute Foundation, Minneapolis, Minnesota, United States

REFERENCES:
- [Result] Traverse JH, McKenna DH, Harvey K, Jorgenso BC, Olson RE, Bostrom N, Kadidlo D, Lesser JR, Jagadeesan V, Garberich R, Henry TD. Results of a phase 1, randomized, double-blind, placebo-controlled trial of bone marrow mononuclear stem cell administration in patients following ST-elevation myocardial infarction. Am Heart J. 2010 Sep;160(3):428-34. doi: 10.1016/j.ahj.2010.06.009. PMID 20826249
- See also: click here for more information on this study — http://www.mplsheart.org